CLINICAL TRIAL: NCT06577181
Title: Effect of Intramuscular Injection of Human Chorionic Gonadotropins on Endometrial Preparation for Frozen Embryo Transfer
Brief Title: Effect of HCG on Endometrial Preparation in Frozen Embryo Transfer
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: Banon fertility center (Unknown)
Responsible Party: Principal Investigator, Omar Ahmed Mohamed Aly Ahmed Nasr, Prof. Ahmed nabil, Assiut University
Other Study IDs: Omar Nasr OBGYN
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: IVF
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women undergoing preparation for Embryo transfer: Group who received intramuscular injection of HCG before embryo transfer
  Interventions: Drug: hCG + estradiol
- Women undergoing preparation for Embryo transfer 1: Group who did not receive intramuscular injection of HCG before embryo transfer
  Interventions: Other: Observation arm

INTERVENTIONS:
Drug: hCG + estradiol — Human chorionic gonadotropins
  Groups: Women undergoing preparation for Embryo transfer
Other: Observation arm — estradiol only wuithout giving hcg
  Groups: Women undergoing preparation for Embryo transfer 1

SUMMARY:
Intramuscular injection of HCG to prepare endometrium for frozen embryo transfer

DETAILED DESCRIPTION:
This study is to compare the effectiveness of intramuscular injections of Human chorionic gonadotropins in preparing the endometrium for frozen embryo transfer compared to the control group who did not receive the injection

ELIGIBILITY:
Inclusion Criteria:

1. Infertile women being prepared for frozen embryo transfer (FET) in an ART program

   Exclusion Criteria:
   * (1) Use of preimplantation genetic test.
2. History of recurrent spontaneous abortion.
3. Presence of congenital uterine malformations.
4. Use of sequential embryo transfer.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Reproductive age female
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy | 2months
  Presence of at least one gestational sac inside the uterus 28 days after embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eftekhar M, Rahmani E, Eftekhar T. Effect of adding human chorionic gonadotropin to the endometrial preparation protocol in frozen embryo transfer cycles. Int J Fertil Steril. 2012 Oct;6(3):175-8. Epub 2012 Dec 17. PMID 24520435